CLINICAL TRIAL: NCT05263973
Title: The Effect of Music on Pain, Comfort and Physiological Parameters During Prematurity: A Randomized Controlled Study
Brief Title: The Effect of Music on Pain, Comfort and Physiological Parameters During Prematurity Retinopathy Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yağmur Sezer Efe, Assist. Prof. Yağmur Sezer Efe, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/122
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: ROP Examination
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Music
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): The infants in the music group (Acem Aşiran Maqam music prepared by TÜMATA group) will be applied music for a about total of 12 minutes, starting 3 minutes before the ROP examination and continuing during the ROP examination, 3 minutes after ROP examination.
  Interventions: Other: Music
- No intervention (No Intervention): The infants in the control group will not be subjected to any intervention other than their clinical routines, only observation will be made.

INTERVENTIONS:
Other: Music — The infants in the music group (Acem Aşiran Maqam music prepared by TÜMATA group) will be applied music for a about total of 12 minutes, starting 3 minutes before the ROP examination and continuing during the ROP examination, 3 minutes after ROP examination
  Arms: Music group

SUMMARY:
It is planned to determine the effect of music during Retinopathy of Prematurity (ROP) examination on pain, comfort and physiological parameters in preterm infants. This is single-center, randomized controlled trial, double blind, parallel.

Hypotheses:

H1: The music applied during the ROP examination has an effect on the Revised Premature Infant Pain Profile (PIPP-R) score of the preterm infant.

H2: The music applied during the ROP examination has an effect on the Preterm Infant Comfort Scale (PMI) score of the preterm infant.

H3: Music applied during the ROP examination has an effect on the physiological parameters (peak heart rate, O2 saturation) of the preterm infant.

H4: The music applied during the ROP examination has an effect on the crying time of the preterm infant during the procedure.

Method: The study will be performed with preterm infants (n=28) hospitalized in the neonatal intensive care unit of a tertiary hospital. Premature infants to be included in the study will be assigned to two study groups using the block randomization method created in the computer environment according to their gestational age, gender, birth weight.

The data in the study were will be collected using the Questionaire Form for Preterm Newborns and Their Parents, Physiological Parameters Observation Form, Revised-Premature Infant Pain Profile (PIPP-R), Premature Infant Comfort Scale (PICS), Pulse Oximeter, Music CD, Music box, Video camera, decibel meter, tripod. Data will be collected by researcher ABÇ. Infants who meet the criteria for inclusion in the study will be selected from the infants who are planned to an ROP examination, and written and verbal consent will be obtained from the families by explaining the purpose of the study.

Questionaire Form for Preterm Newborns and Their Parents will be obtained from the nurse observation form and patient files. Four minutes before the ROP, the infant will be monitored and physiological parameters will be recorded, and three minutes before the ROP, the experimental group will start to listen to music (Video recordings will be evaluated by three experts, PIPP-R and PICS). The music recording will continue to be played during the ROP examination for music group. No application will be made for the control group other than the clinical routines.

DETAILED DESCRIPTION:
This randomized controlled experimental study is planned in order to determine the effect of music on pain, comfort and physiological parameters in preterm infants in ROP examination matched for gestational age, gender and birth weight. The research sample will consist of 28 preterm infants who meet the inclusion criteria. In the literature, the number of infants varies between 10 and 30 in different studies in which music was applied to preterm infants. In this study, it was decided that the number of infants in the groups should be 14 according to α=95% confidence level and 90% power. In the study, it was planned to have 14 infants in the music and control groups. After reaching 28 preterm infants in the study, power analysis will be calculated using pain scores and it will be decided whether the sample size is sufficient or not. All bodies of preterm infants will be recorded with a visible video camera for an average of 10 minutes, 4 minutes before the start of the ROP examination and 4 minutes after the completion of the ROP examination (for PIPP-R and PICS scores). The infants in the music group (Acem Aşiran Maqam music prepared by TÜMATA group) will be applied music for a about total of 10 minutes, starting 3 minutes before the ROP examination and continuing during the ROP examination, 3 minutes after ROP examination. After the necessary disinfection process is done, the voice recorder will be placed in the incubator at a distance of 45 cm from the head of infant and the sound level will be adjusted to an average of 45-60 decibels. The examination will begin with the placement of the speculum in the eye. The duration of the examination varies according to the visibility of the retinal vascularity, and the examination will end with the removal of the speculum from the eye (mean ROP time 1.61 ±1.59). The infants in the control group will not be subjected to any intervention other than their clinical routines, only observation will be made. Data will be collected with the Questionaire Form for Preterm Newborns and Their Parents, Physiological Parameters Observation Form, Revised-Premature Infant Pain Profile (PIPP-R), Premature Infant Comfort Scale (PICS), Pulse Oximeter, Music CD, Music box, Video camera, decibel meter, tripod.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <2000 g,
* Gestational age ≤32 weeks,
* Have not passed the first 2 ROP inspections,
* Not receiving ventilatory support (not intubated or positive pressure ventilation support) for the last 72 hours,
* Vital signs within normal limits (without tachycardia, tachypnea, hyperthermia, hypothermia, dyspnea, intercostal or subcostal retraction),
* Not having any congenital anomalies (eye, neurological) that may adversely affect the examination,
* No hearing problem,
* No painful intervention is performed at least 30 minutes before the ROP examination,
* Preterm newborns whose corrected/postnatal age is 28-36 weeks at the time of examination,
* Newborns whose mothers want to participate in the study will be included in the study.

Exclusion Criteria:

* Clinic condition worsening during working,
* Diagnosed with hydrocephalus, necrotizing enterocolitis, indirect hyperbilirubinemia,
* Receiving analgesic treatment,
* Newborns whose mothers want to withdraw from the study will be excluded from the study groups.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Premature Infant Comfort Scale (PBIC) | The measurement will start 4 minutes before the ROP examination and will end 4 minutes after the ROP examination.
  According to the PICS, a score between 7-35 is obtained from the scale. A high score from the scale indicates a low level of comfort.
Premature Baby Pain Profile Scale-Revised Form (PIPP-R) | The measurement will start 4 minutes before the ROP examination and will end 4 minutes after the ROP examination.
  The PIPP-R is a Likert-type scale. In scoring the scale, items related to physiological and behavioral elements are scored as 0, 1, 2, 3, reflecting the difference between the values at baseline and during the procedure in each variable. Contextual items (behavioral status and CI) are scored as 3, 2, 1, 0 only at the beginning of the pain assessment (before touching the baby). According to the PIPP-R, the baby's pain is evaluated over the total score. Accordingly, the highest score that can be obtained from the PIPP-R scale for preterm newborns is 21 and 18 for term newborns.
Physiological parameters- heart rate | The measurement will start 4 minutes before the ROP examination and will end 4 minutes after the ROP examination.
  Heart rate
Physiological parameters- oxygen saturation | The measurement will start 4 minutes before the ROP examination and will end 4 minutes after the ROP examination.
  Oxygen saturation
Physiological parameters- respiratory rate | The measurement will start 4 minutes before the ROP examination and will end 4 minutes after the ROP examination.
  Respiratory rate
Physiological parameters- crying time | immediately after the ROP examination.
  Crying time

CONTACTS AND LOCATIONS:
Overall Officials: Yağmur Sezer Efe, Assist. Prof., Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes university, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Cuhaci AB, Efe YS, Gunes T. The effect of music on pain, comfort, and physiological parameters during premature retinopathy examination. J Pediatr Nurs. 2024 Sep-Oct;78:149-157. doi: 10.1016/j.pedn.2024.06.020. Epub 2024 Jun 28. PMID 38943838